CLINICAL TRIAL: NCT00083629
Title: PET Whole Body Biodistribution and Test Retest Brain Imaging Studies Using a Dopamine Transporter Ligand [18F]FECNT
Brief Title: Use of [18F]FECNT in Positron Emission Tomography
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Mental Health (NIMH) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 040204; 04-M-0204
Record Dates: First submitted 2004-05-27; First posted 2004-05-27 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2005-09

CONDITIONS: Healthy
Keywords: [18F]FECNT; Biodistribution; Dosimetry; Dopamine Transporter; MIRD; Kinetic Analysis; Compartment Analysis; Healthy Volunteer; HV

INTERVENTIONS:
Procedure: PET

SUMMARY:
This study will examine the use of a new radioactive tracer called [18F]FECNT in positron emission tomography (PET) scanning for measuring dopamine transporter (DAT) in the brain. DAT is found in brain neurons (nerve cells) that release the chemical messenger dopamine. By taking pictures of the DAT, scientists hope to learn more about the function of these neurons.

Normal, healthy volunteers between 18 and 65 years of age may be eligible for this study. Candidates are screened with a medical history and physical examination, psychological assessment, and blood and urine tests.

Subjects enrolled in the study participate in one of the following procedures:

Brain Imaging Study: Part 1

Two catheters (small plastic tubes) are placed into veins in the subject's arms for injecting [18F]FECNT and for collecting blood samples during the scan. A third catheter is placed into a wrist artery to obtain arterial blood during the scan. With the catheters in place, the subject lies down on the scanner bed with his or her head placed in a special mask that limits movement during the brain scan. The scan begins with an initial x-ray like picture for about 10 minutes, after which the [18F]FECNT is injected and the actual PET scan starts. The entire procedure takes about 6 hours, including 2 hours of continuous scanning sessions, during which the subject is required to lie still. Subjects can relax out of the scanner between scans. They are monitored throughout the procedure. Vital signs are measured and electrocardiogram is taken once before and twice after injection of the tracer. At the end of the scanning, additional blood and urine samples are collected. Subjects are asked to urinate every 2 hours to lessen the radioactivity in the body.

Whole Body Imaging Study: Part 2

For this procedure, a catheter is placed in a vein for injecting the [18F]FECNT tracer. A total of five scans are taken, each one spanning from head to upper thigh. During the course of the scans, x-ray like pictures are obtained. The first scan takes about 100 minutes. Four additional 1-hour scans are done every 100 minutes. The total time for the scans is about 6 hours, and the total time for the entire procedure is about 9 hours. About 2 tablespoons of blood are drawn by needle stick at one time during the imaging. Subjects can leave the PET scanner between scans. They are asked to urinate every 2 hours for 6 hours from the time of tracer injection and to collect all the urine so that radioactivity can be measured.

Brain Imaging Study: Part 3

Part 3 of the study is the same as Part 1, except that two PET procedures are done on separate days, the second within 4 weeks of the first. In addition, participants may also under magnetic resonance imaging (MRI) scanning, a test that uses magnetic fields and radio waves to obtain pictures of the brain.

DETAILED DESCRIPTION:
The dopamine system plays important roles in various neurological and psychiatric disorders such as Parkinson's disease, schizophrenia, mood disorders, and attention-deficit hyperactivity disorder. Several positron emission tomography (PET) and single photon emission computed topography (SPECT) tracers have been developed including [11C]CFT and [123I]beta-CIT. These tracers have been successfully applied in patients, particularly to stage those with Parkinson's disease. However, these tracers lack selectivity among monoamine (dopamine, serotonin, and norepinephrine) transporters. Recently a new PET tracer, [18F]FECNT brain uptake and washout has been developed, which has high selectivity and affinity to the dopamine transporter (DAT). Part 1 of this study will measure the kinetics of [18F]FECNT brain uptake and washout. Part 2 will estimate radiation-absorbed doses in healthy human subjects by performing whole body PET imaging studies. Part 3 will assess the reliability of measuring DAT densities in the brain by performing a test retest brain PET studies in healthy human subjects. The results of this overall study are required to apply this tracer in various neurological and psychiatric disorders in the future.

ELIGIBILITY:
INCLUSION CRITERIA:

Healthy subjects ages 18-65

EXCLUSION CRITERIA-WHOLE BODY IMAGING:

Current diagnosis of psychiatric disease, substance dependence or severe systemic disease.

History of substance abuse within 6 months.

Abnormal laboratory tests.

Prior participation in other research protocols within the past year such that a radiation exposure together with the present study would exceed the annual limits.

Pregnancy and breast feeding.

HIV positive.

EXCLUSION CRITERIA-DYNAMIC BRAIN IMAGING:

Current diagnosis of psychiatric disease, substance dependence or severe systemic disease.

History of substance abuse within 6 months.

Abnormal laboratory tests.

Novocain allergy.

Prior participation in other research protocols within the past year such that a radiation exposure together with the present study would exceed the annual limits.

Any condition that increases increase risk for MRI (e.g., pacemaker, metallic foreign body in the eye).

Pregnancy and breast feeding.

HIV positive.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2004-05; Study Completion 2005-09

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Mental Health (NIMH), Bethesda, Maryland, United States

REFERENCES:
- [Background] Abi-Dargham A, Gandelman M, Zoghbi SS, Laruelle M, Baldwin RM, Randall P, Zea-Ponce Y, Charney DS, Hoffer PB, Innis RB. Reproducibility of SPECT measurement of benzodiazepine receptors in human brain with iodine-123-iomazenil. J Nucl Med. 1995 Feb;36(2):167-75. PMID 7830108
- [Background] Barrio JR, Huang SC, Melega WP, Yu DC, Hoffman JM, Schneider JS, Satyamurthy N, Mazziotta JC, Phelps ME. 6-[18F]fluoro-L-dopa probes dopamine turnover rates in central dopaminergic structures. J Neurosci Res. 1990 Dec;27(4):487-93. doi: 10.1002/jnr.490270408. PMID 2127807
- [Background] Cloutier RJ, Smith SA, Watson EE, Snyder WS, Warner GG. Dose to the fetus from radionuclides in the bladder. Health Phys. 1973 Aug;25(2):147-61. doi: 10.1097/00004032-197308000-00009. No abstract available. PMID 4784245